CLINICAL TRIAL: NCT06452849
Title: Temporal Interference Stimulation of Amygdala and dLPFC: A Randomized Controlled Trial for Adolescent Depression
Brief Title: Amygdala and dLPFC MRI-TIS for Depression in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pudong New Area Mental Health Center, School of Medicine, Tongji University (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, huangjingjing, Chief Physician, Shanghai Pudong New Area Mental Health Center, School of Medicine, Tongji University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDJW-2024-001CSB
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
Keywords: Adolescents; Deep Brain Stimulation; Major Depressive Disorder; Temporal Interference; Amygdala
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amygdala TI (Experimental): Right amygdala Temporal Interference (TI) stimulation with 100 frequency difference, 20 minutes per day for 5 days.
  Interventions: Device: Nervio-X
- dLPFC TI (Experimental): L_dLPFC TI Temporal Interference (TI) stimulation with 10 frequency difference, 20 minutes per day for 5 days.
  Interventions: Device: Nervio-X

INTERVENTIONS:
Device: Nervio-X — An 8-channel TIS device developed by NEURODOME Corporation.

SUMMARY:
The study utilizes a non-invasive deep brain stimulation (temporal interference, TI) technique primarily targeting the amygdala to preliminarily explore the clinical efficacy and potential mechanisms of MRI-compatible TI technology in regulating the amygdala in adolescent depressive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged between 14 and 18, with no gender restrictions;
* A diagnosis of depression made by the study physician based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
* HAMD-17 score of 17 or higher;
* Participants must not have changed their antidepressant medication regimen from 30 days prior to signing the informed consent form through the duration of the experiment;
* Eligible individuals or their authorized representatives must demonstrate, as assessed by the study physician, a comprehensive understanding of the study's objectives and procedures, be capable of adhering to the requirements set forth in the study protocol, and provide their signature on the informed consent form.

Exclusion Criteria:

* Eligible participants must not have a history of psychiatric or neurological disorders, as judged by the investigator, which may impact the evaluation of the study's efficacy;
* Participants must not have a history of seizures or prior episodes of epilepsy;
* The presence of metallic foreign objects within the cranial structure or metallic cardiac implants;
* Participants must not have a diagnosis of organic brain disease, nor a history of significant cranial trauma or neurosurgical intervention;
* Participants received electroconvulsive therapy or other physical therapies (such as transcranial magnetic stimulation therapy); The researcher evaluated the individual's mental state and determined it to present a significant risk of suicidal ideation or behavior;
* Pregnant or breastfeeding;
* Participants who are concurrently engaged in other clinical interventional trials;
* Participants presenting with other circumstances that the investigator deems unsuitable for the intervention being studied

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
HAMD-17 | Baseline, after treatment, 1 week, 4 weeks and 8 weeks
HAMA | Baseline, after treatment, 1 week, 4 weeks and 8 weeks
MADRS | Baseline, after treatment, 1 week, 4 weeks and 8 weeks
PHQ-A | Baseline, after treatment, 1 week, 4 weeks and 8 weeks
GAD-7 | Baseline, after treatment, 1 week, 4 weeks and 8 weeks
SHAPS | Baseline, 4 weeks and 8 weeks
PSQI | Baseline, 4 weeks and 8 weeks
SF-36 | Baseline and 8 weeks
WHOQOL-BREF | Baseline and 8 weeks
ARI | Baseline and 8 weeks
OSI | Baseline, 4 weeks and 8 weeks
  For use when the patient exhibits self-harming behavior

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pudong New Area Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No